CLINICAL TRIAL: NCT01165554
Title: A Principal Open-Label Study to Compare the Brain Uptake of [18F]Flutemetamol With Brain Amyloid Levels Determined Post-Mortem
Brief Title: Positron Emission Tomography (PET) Imaging of Brain Amyloid Compared to Post-Mortem Levels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: i3 Statprobe (Industry); Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-067-007
Record Dates: First submitted 2010-06-21; First posted 2010-07-20 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Brain Fibrillarab Levels
Keywords: Amyloid; PET-Positron Emission Tomography; SUVR-Standard uptake value ratios
MeSH Terms: conditions — Alzheimer Disease | interventions — flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F] Flutemetamol (Experimental)
  Interventions: Drug: [18F] Flutemetamol

INTERVENTIONS:
Drug: [18F] Flutemetamol — Flutemetamol (18F) Injection, 111 to 370 MBq (3 to 10 mCi), single intravenous injection.
  Other Names: AH110690

SUMMARY:
To determine the level of association between quantitative regional estimates of brain uptake of [18F]flutemetamol and quantitative immunohistochemical regional estimates of brain levels of amyloid estimated from post-mortem analysis of corresponding brain tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a short life expectancy (approximately 1 year or less) as estimated by the Investigator.
* The subject is 70 years of age or older if cognitively normal, or 55 years of age or older if terminal because of dementia.
* The subject's general health is adequate to undergo the study procedures.

Exclusion Criteria:

* The subject has a contraindication for PET.
* The subject has a known or suspected hypersensitivity/allergy to [18F]flutemetamol or to any of the excipients.
* The subject is unable to tolerate or cooperate with study procedures.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sherwin, MD, PhD, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

REFERENCES:
- [Derived] Kim SJ, Jang H, Yoo H, Na DL, Ham H, Kim HJ, Kim JP, Farrar G, Moon SH, Seo SW. Clinical and Pathological Validation of CT-Based Regional Harmonization Methods of Amyloid PET. Clin Nucl Med. 2024 Jan 1;49(1):1-8. doi: 10.1097/RLU.0000000000004937. Epub 2023 Nov 29. PMID 38048354
- [Derived] Tome SO, Tsaka G, Ronisz A, Ospitalieri S, Gawor K, Gomes LA, Otto M, von Arnim CAF, Van Damme P, Van Den Bosch L, Ghebremedhin E, Laureyssen C, Sleegers K, Vandenberghe R, Rousseau F, Schymkowitz J, Thal DR. TDP-43 pathology is associated with increased tau burdens and seeding. Mol Neurodegener. 2023 Sep 30;18(1):71. doi: 10.1186/s13024-023-00653-0. PMID 37777806
- [Derived] Thal DR, Ronisz A, Tousseyn T, Rijal Upadhaya A, Balakrishnan K, Vandenberghe R, Vandenbulcke M, von Arnim CAF, Otto M, Beach TG, Lilja J, Heurling K, Chakrabarty A, Ismail A, Buckley C, Smith APL, Kumar S, Farrar G, Walter J. Different aspects of Alzheimer's disease-related amyloid beta-peptide pathology and their relationship to amyloid positron emission tomography imaging and dementia. Acta Neuropathol Commun. 2019 Nov 14;7(1):178. doi: 10.1186/s40478-019-0837-9. PMID 31727169
- [Derived] Thal DR, Beach TG, Zanette M, Lilja J, Heurling K, Chakrabarty A, Ismail A, Farrar G, Buckley C, Smith APL. Estimation of amyloid distribution by [18F]flutemetamol PET predicts the neuropathological phase of amyloid beta-protein deposition. Acta Neuropathol. 2018 Oct;136(4):557-567. doi: 10.1007/s00401-018-1897-9. Epub 2018 Aug 19. PMID 30123935
- [Derived] Ikonomovic MD, Buckley CJ, Heurling K, Sherwin P, Jones PA, Zanette M, Mathis CA, Klunk WE, Chakrabarty A, Ironside J, Ismail A, Smith C, Thal DR, Beach TG, Farrar G, Smith AP. Post-mortem histopathology underlying beta-amyloid PET imaging following flutemetamol F 18 injection. Acta Neuropathol Commun. 2016 Dec 12;4(1):130. doi: 10.1186/s40478-016-0399-z. PMID 27955679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started on May, 2010 and ended on November 2011.
Pre-assignment Details: 23 subjects withdrew from study prior to dosing of the product.
Groups:
- Flutemetamol Injection: [18F]flutemetamol (less than 10 microgram (ug) flutemetamol). The nominal activity of a single administration of [18F]flutemetamol was 185 to 370 megabecquerels (MBq).
Period: Overall Study
Arm/Group | Flutemetamol Injection
Started | 203 (This was the number of subjects that started the study.)
Completed | 180
Not Completed | 23
Not completed — Withdrawal by Subject | 23

BASELINE CHARACTERISTICS:
Arm/Group | Flutemetamol Injection
Number analyzed (Participants) | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 165
Age Continuous [Mean (Standard Deviation); unit: years] | 79.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 77
Region of Enrollment [Number; unit: participants]
  United States | 168
  United Kingdom | 12

OUTCOME MEASURES:

1. Primary Outcome: The Sensitivity of Blinded Visual Interpretations of [18F]Flutemetamol Positron Emission Tomography (PET) Images Without Anatomic Brain Images for Detecting Brain Fibrillar Amyloid β.
Description: A calculation used to assess Sensitivity was (Number of Blinded Reads determined abnormal by Reader "N") divided by the (Total number of abnormal participants).
  Blinded visual interpretations of [18F]flutemetamol Positron Emission Tomography (PET) images without anatomic brain images for detecting brain fibrillar amyloid β.
Time Frame: Post flutemetamol administration.
Population: The assessments were post-mortum based on the estimates of the presence of amyloid plaque in the brain.
Measure: Number; unit: Percentage of Sensitivity by Reader
Arm/Group | Sensitivity Percentage of Abnormal Visual Reads
Number analyzed (Participants) | 43
Percentage of Sensitivity by Reader
  Reader 1- Abnormal | 81
  Reader 2 - Abnormal | 88
  Reader 3 - Abnormal | 93
  Reader 4 - Abnormal | 93
  Reader 5 - Abnormal | 88

2. Secondary Outcome: Blinded Visual Interpretation of Each Subject's Flutemetamol F 18 Injection Brain PET Images as Normal, Without Anatomic Brain Images.
Description: A calculation used to assess Specificity was (Number of Blinded Reads determined normal by Reader "N") divided by the (Total number of normal participants).
  Blinded visual interpretation of each subject's Flutemetamol F 18 Injection brain PET images as normal, without anatomic brain images.
Time Frame: Post Flutemetamol administrations
Population: The assessment was done post-mortum based on the estimates of the presence of amyloid plaque in the brain.
Measure: Number; unit: Percentage of Specificity by Reader
Arm/Group | Specificity Percentage of Normal Visual Reads
Number analyzed (Participants) | 25
Percentage of Specificity by Reader
  Reader 1 - Normal | 88
  Reader 2 - Normal | 92
  Reader 3 - Normal | 44
  Reader 4 - Normal | 80
  Reader 5 - Normal | 92

3. Secondary Outcome: Blinded Visual Interpretation of Each Subject's Flutemetamol F 18 Injection Brain PET Images as Abnormal, With Anatomic CT Brain Images for Reference.
Description: Blinded visual interpretation of each subject's Flutemetamol F 18 Injection brain PET images as abnormal, with anatomic CT brain images for reference.
Time Frame: Post flutemetamol administration.
Measure: Number (95% Confidence Interval); unit: Percent of Sensitivity-Abnormal Reads
Groups:
- Sensitivity-Abnormal Visual Reads: [18F]flutemetamol (less than 10 microgram (ug) flutemetamol). The nominal activity of a single administration of [18F]flutemetamol was 185 to 370 megabecquerels (MBq).
Arm/Group | Sensitivity-Abnormal Visual Reads
Number analyzed (Participants) | 43
Percent of Sensitivity-Abnormal Reads
  Reader 1 | 91 [78 to 97]
  Reader 2 | 95 [84 to 99]
  Reader 3 | 98 [88 to 100]
  Reader 4 | 91 [78 to 97]
  Reader 5 | 91 [77 to 97]

4. Secondary Outcome: Blinded Visual Interpretation of Each Subject's Flutemetamol F 18 Injection Brain PET Images as Normal, With Anatomic CT Brain Images for Reference.
Description: Blinded visual interpretation of each subject's Flutemetamol F 18 Injection brain PET images as normal, with anatomic CT brain images for reference.
Time Frame: Post flutemetamol administration.
Measure: Number (95% Confidence Interval); unit: Percent of Specificity-Normal Reads
Groups:
- Specificity-Normal Visual Reads: [18F]flutemetamol (less than 10 microgram (ug) flutemetamol). The nominal activity of a single administration of [18F]flutemetamol was 185 to 370 megabecquerels (MBq).
Arm/Group | Specificity-Normal Visual Reads
Number analyzed (Participants) | 25
Percent of Specificity-Normal Reads
  Reader 1 | 92 [74 to 99]
  Reader 2 | 88 [69 to 98]
  Reader 3 | 56 [35 to 76]
  Reader 4 | 88 [69 to 98]
  Reader 5 | 92 [74 to 99]

ADVERSE EVENTS:
Arm/Group | Flutemetamol Injection
Serious Adverse Events (participants affected / at risk) | 4/180
Other Adverse Events (participants affected / at risk) | 0/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flutemetamol Injection (N=180)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Senile Dementia (Psychiatric disorders) | 1 (1)
Change in Mental Status (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No